CLINICAL TRIAL: NCT04573517
Title: Early Amniotomy Following Transcervical Foley Balloon in the Induction of Labor: a Randomized Clinical Trial
Brief Title: Early Amniotomy Following Transcervical Foley Balloon in the Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0163
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Labor Induction; Early Amniotomy
Keywords: Foley balloon
MeSH Terms: interventions — Amniotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early amniotomy (Experimental): Subjects randomized to this arm will undergo amniotomy within 2 hours of removal of Foley balloon.
  Interventions: Procedure: Amniotomy; Device: Foley balloon
- Delayed amniotomy (Active Comparator): Subjects randomized to this arm will undergo amniotomy at least 4 hours after removal of Foley balloon.
  Interventions: Procedure: Amniotomy; Device: Foley balloon

INTERVENTIONS:
Procedure: Amniotomy — Artificial rupture of amniotic membranes
Device: Foley balloon — The Foley balloon is inserted transcervically and inflated to a volume of 60 cc. It may be spontaneously expelled or manually removed if in place for 12 hours.
  Other Names: Foley catheter; Foley bulb

SUMMARY:
Amniotomy is commonly done in the management of labor, though there is little research guiding the timing of amniotomy. Recent research largely suggests a benefit to earlier amniotomy, reporting shorter labor courses with no increase in the number of cesarean deliveries. This is some research, however, that reports an increase in cesarean deliveries with early amniotomy. Due to the small number of studies evaluating this topic, as well as the conflicting results, more research is needed. Additionally, the method of cervical ripening prior to amniotomy should be accounted for, as it may have an impact on the overall labor course. The purpose of this study is to evaluate the impact of early versus delayed amniotomy on time of delivery time from induction to the active phase of labor, as well on total time to delivery and maternal and neonatal outcomes in women undergoing cervical ripening with the Foley balloon.

DETAILED DESCRIPTION:
This will be an unblinded randomized clinical trial. The investigators will recruit 174 pregnant women undergoing induction of labor. Recruitment will occur on the Labor and Delivery unit at the time of induction, after the decision has been made to place a Foley balloon for cervical ripening. Enrolled subjects will be randomized to early or delayed amniotomy.

Subjects randomized to early amniotomy will undergo amniotomy within 2 hours of Foley balloon removal. Subjects randomized to delayed amniotomy will undergo amniotomy at least 4 hours after Foley balloon removal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18
* Singleton pregnancy
* Term gestation (37 weeks gestation)
* Cephalic presentation
* Undergoing labor induction with transcervical Foley balloon

Exclusion Criteria:

* Previous uterine surgery
* Prelabor rupture of membranes
* Severe pre-eclampsia, HELLP, or eclampsia
* HIV, HCV, or HBV
* Heart disease
* Fever (≥38 0C) at admission
* Category II or III fetal heart rate tracing prior to randomization
* Polyhydramnios
* Fetal growth restriction <3%
* EFW > 4200 g
* Fetal demise or major congenital anomaly
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Berry, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Berry M, Lamiman K, Slan MN, Zhang X, Arena Goncharov DD, Hwang YP, Rogers JA, Pacheco LD, Saade GR, Saad AF. Early vs delayed amniotomy following transcervical Foley balloon in the induction of labor: a randomized clinical trial. Am J Obstet Gynecol. 2024 May;230(5):567.e1-567.e11. doi: 10.1016/j.ajog.2024.01.028. Epub 2024 Feb 15. PMID 38367749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 subjects were enrolled between October 2020 and March 2023.
Period: Overall Study
Arm/Group | Early Amniotomy | Delayed Amniotomy
Started | 75 | 75
Completed | 75 | 74
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were excluded after enrollment but prior to assignment to groups. However, one participant was excluded after group assignment but prior to the intervention due to the development of a contraindication to the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Amniotomy | Delayed Amniotomy | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 74 | 149
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 24 [18 to 43] | 24 [18 to 40] | 24 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 60 | 61 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Active Phase of Labor
Description: Total time from initiation of labor induction to reaching 6 cm cervical dilation
Time Frame: At delivery
Measure: Median (Full Range); unit: minutes
Arm/Group | Early Amniotomy | Delayed Amniotomy
Number analyzed (Participants) | 75 | 74
minutes | 885 [161 to 2340] | 975 [250 to 2760]

2. Secondary Outcome: Time to Delivery
Description: Total time from initiation of labor induction to delivery
Time Frame: At delivery
Reporting Status: Not Posted

3. Secondary Outcome: Vaginal Delivery Rate
Description: Rate of vaginal delivery within 24, 36, and 48 hours
Time Frame: At delivery
Reporting Status: Not Posted

4. Secondary Outcome: Cesarean Section Rate
Description: Rate of cesarean section and indications
Time Frame: At delivery
Reporting Status: Not Posted

5. Secondary Outcome: Maternal Infection Composite
Description: Includes isolated maternal fever, chorioamnionitis, endometritis, wound infection
Time Frame: From admission to discharge, up to 2 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Umbilical Cord Prolapse
Description: Rates of umbilical cord prolapse
Time Frame: At delivery
Reporting Status: Not Posted

7. Secondary Outcome: Neonatal Outcome Composite
Description: Neonatal outcome composite including NICU admission, respiratory support, hypoxic ischemic encephalopathy, seizures, sepsis, meconium aspiration syndrome, birth trauma, intracranial or subgaleal hemorrhage, hypotension requiring pressors, and perinatal death.
Time Frame: From admission to discharge, up to 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Until the time of discharge from the hospital, an average of 3 days
Arm/Group | Early Amniotomy | Delayed Amniotomy
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 0/75 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04573517/Prot_SAP_000.pdf